CLINICAL TRIAL: NCT02654847
Title: Norepinephrine To Prevent Hypotension After Spinal Anesthesia For Cesarean Delivery: A Dose Finding Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-02
Record Dates: First submitted 2016-01-05; First posted 2016-01-13 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Hypotension
Keywords: vasopressor; blood pressure; Cesarean section; spinal anesthesia
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Norepinephrine 3 micrograms/mL (Active Comparator): 1mL of a solution of norepinephrine, containing 3 micrograms/mL in normal saline, will be given intravenously to a patient if her blood pressure decreases from baseline.
  Interventions: Drug: Norepinephrine; Drug: Normal Saline
- Norepinephrine 4 micrograms/mL (Active Comparator): 1mL of a solution of norepinephrine, containing 4 micrograms/mL in normal saline, will be given intravenously to a patient if her blood pressure decreases from baseline.
  Interventions: Drug: Norepinephrine; Drug: Normal Saline
- Norepinephrine 5 micrograms/mL (Active Comparator): 1mL of a solution of norepinephrine, containing 5 micrograms/mL in normal saline, will be given intravenously to a patient if her blood pressure decreases from baseline.
  Interventions: Drug: Norepinephrine; Drug: Normal Saline
- Norepinephrine 6 micrograms/mL (Active Comparator): 1mL of a solution of norepinephrine, containing 6 micrograms/mL in normal saline, will be given intravenously to a patient if her blood pressure decreases from baseline.
  Interventions: Drug: Norepinephrine; Drug: Normal Saline
- Norepinephrine 7 micrograms/mL (Active Comparator): 1mL of a solution of norepinephrine, containing 7 micrograms/mL in normal saline, will be given intravenously to a patient if her blood pressure decreases from baseline.
  Interventions: Drug: Norepinephrine; Drug: Normal Saline
- Norepinephrine 8 micrograms/mL (Active Comparator): 1mL of a solution of norepinephrine, containing 8 micrograms/mL in normal saline, will be given intravenously to a patient if her blood pressure decreases from baseline.
  Interventions: Drug: Norepinephrine; Drug: Normal Saline

INTERVENTIONS:
Drug: Norepinephrine
  Other Names: Norepinephrine bitartrate
Drug: Normal Saline — 0.9% sodium chloride solution, used as a diluent.
  Other Names: sodium chloride

SUMMARY:
Spinal anesthesia is the most common anesthetic technique for elective Cesarean delivery (CD), but the most frequent unwanted side effect is hypotension, which can cause nausea and vomiting, as well as effects on the fetus. Prevention and treatment of maternal hypotension includes intravenous fluids and vasopressors. Phenylephrine is the most common vasopressor used for this purpose. However, it has been shown to reduce maternal heart rate and cardiac output, which may be a concern in an already compromised fetus. Norepinephrine is commonly used in high concentrations in intensive care and recent studies have suggested that in low concentrations it may be a better alternative to phenylephrine in elective CD, as it does not reduce the maternal heart rate or cardiac output. The optimum bolus dose of norepinephrine to prevent hypotension after spinal anesthesia in elective CD has not been elucidated. The investigators propose this study to determine the dose that would be effective in 90% of patients (ED90).

A previous study by Ngan Kee et al, using continuous infusion of norepinephrine to prevent hypotension in elective CD, suggested a potency ratio for norepinephrine to phenylephrine of approximately 16:1. Hence, the investigators hypothesise that the ED90 will be approximately 6 µg, given that the current phenylephrine bolus dose at the investigators' institution is approximately 100 µg.

DETAILED DESCRIPTION:
The use of norepinephrine to prevent and treat hypotension during cesarean delivery (CD) is new and data in the literature are scarce. A recent randomised controlled trial by Ngan Kee et al compared continuous infusions of norepinephrine and phenylephrine to prevent hypotension during CD. They showed that norepinephrine was effective at maintaining blood pressure, with a greater cardiac output and heart rate compared to phenylephrine. However, the effective bolus dose of norepinephrine needed to prevent maternal hypotension was not determined, and since this is a relatively new arena, no dose-response studies are available in the literature either. Therefore, it would be logical to establish the effective bolus dose of norepinephrine TO PREVENT HYPOTENSION during elective CD.

ELIGIBILITY:
Inclusion Criteria:

* Elective CD under spinal anesthesia
* Normal singleton pregnancy beyond 36 weeks gestation
* ASA physical status II/III
* Weight 50-100 kg, height 150-180 cm
* Age over 18 years
* Informed consent

Exclusion Criteria:

* Patient refusal
* Allergy or hypersensitivity to norepinephrine or sulfite
* Preexisting or pregnancy-induced hypertension
* Cardiovascular or cerebrovascular disease
* Fetal abnormalities
* History of diabetes, excluding gestational diabetes
* Use of monoamine oxidase inhibitors, triptyline or imipramine antidepressants

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 30 minutes
  The primary outcome of this study will be the success/response of the norepinephrine dose to maintain the systolic blood pressure at or above 80% of baseline, from induction of spinal anesthesia to delivery of the fetus.

SECONDARY OUTCOMES:
Presence of Nausea | 30 minutes
  Presence of nausea in patients from induction of spinal anesthesia to delivery of the fetus.
Presence of Vomiting | 30 minutes
  Presence of vomiting in patients from induction of spinal anesthesia to delivery of the fetus.
Hypertension: Systolic blood pressure at or above 120% of baseline | 30 minutes
  Systolic blood pressure at or above 120% of baseline, from induction of spinal anesthesia to delivery of the fetus.
Bradycardia: Heart rate less than 50 bpm | 30 minutes
  Heart rate less than 50 bpm, from induction of spinal anesthesia
Upper sensory level of anesthetic block, assessed by pinprick upon delivery | 30 minutes
  Upper sensory level of anesthesia, assessed by pinprick upon delivery
Umbilical artery pH | 24 hours
  Umbilical artery pH
Umbilical artery partial pressure of carbon dioxide | 24 hours
  Umbilical artery partial pressure of carbon dioxide
Umbilical artery partial pressure of oxygen | 24 hours
  Umbilical artery partial pressure of oxygen
Umbilical artery bicarbonate | 24 hours
  Umbilical artery bicarbonate
Umbilical artery base excess | 24 hours
  Umbilical artery base excess
Umbilical vein pH | 24 hours
  Umbilical vein pH
Umbilical vein partial pressure of carbon dioxide | 24 hours
  Umbilical vein partial pressure of carbon dioxide
Umbilical vein partial pressure of oxygen | 24 hours
  Umbilical vein partial pressure of oxygen
Umbilical vein bicarbonate | 24 hours
  Umbilical vein bicarbonate
Umbilical vein base excess | 24 hours
  Umbilical vein base excess

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Onwochei DN, Ngan Kee WD, Fung L, Downey K, Ye XY, Carvalho JCA. Norepinephrine Intermittent Intravenous Boluses to Prevent Hypotension During Spinal Anesthesia for Cesarean Delivery: A Sequential Allocation Dose-Finding Study. Anesth Analg. 2017 Jul;125(1):212-218. doi: 10.1213/ANE.0000000000001846. PMID 28248702